CLINICAL TRIAL: NCT06175091
Title: Impact of an Alarm Management Protocol on Noise Pollution and Patient Safety in Intensive Care Units
Acronym: REALARM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20PH287; ANSM (Other: 2022-A00454-39)
Record Dates: First submitted 2023-11-20; First posted 2023-12-18 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Intensive Care Unit
Keywords: alarm fatigue; nursing staff; Resuscitation patients; restrictive alarm strategy
MeSH Terms: conditions — Alert Fatigue, Health Personnel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Usual management, i.e. alarm management left to the discretion of the nurse caring for the patient.
  Interventions: Device: alarm management left to the discretion of the nurse
- intervention group (Experimental): restrictive alarm strategy
  Interventions: Device: restrictive alarm use strategy

INTERVENTIONS:
Device: alarm management left to the discretion of the nurse — alarm management left to the discretion of the nurse in charge of the patient
  Arms: control group
Device: restrictive alarm use strategy — more restrictive protocol for the use of alarms
  Arms: intervention group

SUMMARY:
Resuscitation patients are monitored for various physiological parameters. When these parameters exceed abnormal thresholds, an audible alarm is triggered. Given the complexity of physiological situations and the number of monitored parameters, the number of alarms within an intensive care unit is significant. In the literature, the number ranges from 100 to 350 alarms per patient per day. Among these alarms, 74 to 99% are deemed irrelevant as they provide false or insignificant information. This study will enable to assess the efficacy of a restrictive protocol for managing alarms as a means of rationalizing their use.

DETAILED DESCRIPTION:
The large volume of unnecessary alarms has multiple negative repercussions. Firstly, the excessively loud sound environment present in most resuscitation services causes stress and discomfort for both patients and caregivers. Additionally, nurses become desensitised and less responsive when the number of alarms is high, particularly if many of them are ultimately pointless. Finally, multiple interruptions of tasks associated with alarms that require responses are sources of errors in the execution of care and medication preparation.

These interruptions contribute to a phenomenon known as "alarm fatigue", which many authorsand health authorities consider a threat to patient safety.The intensive care unit of the Saint-Etienne University Hospital has had a long-standing interest in this topic, and has a computerized data collection tool that permits exhaustive analysis of all alarm signals originating from each resuscitation bed.

This study will enable to assess the efficacy of a restrictive protocol for managing alarms as a means of rationalizing their use.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* Patient admitted to the intensive care unit of the ST-ETIENNE University Hospital
* Patient affiliated or entitled to a social security system
* Patient having received informed information about the study and having co-signed, with the investigator, a consent to participate in the study or, for patients who are unable to consent due to health condition, a trusted person/family member who has been informed about the study and has who has co-signed, with the investigator, a consent to participate

Exclusion Criteria:

* Pregnant and nursing women
* Persons of legal age under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
efficiency criterion: the number of alarms per patient per day | 1 month
  An efficiency criterion: the number of alarms per patient per day
A safety criterion: the length of time patients have potentially dangerous heart rate, blood pressure or oxygen saturation values | 1 month
  A safety criterion: the length of time patients have potentially dangerous heart rate, blood pressure or oxygen saturation values.

SECONDARY OUTCOMES:
Incidence of serious adverse events | 1 month
  Incidence of serious adverse events
Alarm response time | 1 month
  Alarm response time: the time between the alarm being triggered and the acoustic signal being silenc
Evaluation of patient perception using the Discomforts of intensive care patients questionnaire | 1 month
  Evaluation of patient perception using the Discomforts of intensive care patients questionnaire. The Discomforts of intensive care patients questionnaire validated in intensive care and in French, assesses 16 sources of discomfort, including noise. The questionnaire is given to patients before they are discharged from intensive care. The questionnaire scores range from 0 to 100, with the highest score indicating maximum discomfort.
Sound level measurement using a sound level meter | 7 days
  Sound level measurement using a sound level meter. A measuring instrument will be placed in the rooms of the patients included during the day for 4 consecutive hours on day 1, 3 and 7. This part of the study will be carried out in conjunction with occupational medicine and the Quality, Risk Management and Patient Experience Department, which already carry out this type of measurement as part of their assessment of working conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Thiéry, PhD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France